CLINICAL TRIAL: NCT02254733
Title: Enhancing Assertive Community Treatment With Cognitive Behavioral Therapy and Social Skills Training for Schizophrenia.
Brief Title: Assertive Community Treatment With CBT and SST for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01MH091057 (NIH); 5R01MH091057 (NIH)
Record Dates: First submitted 2014-04-25; First posted 2014-10-02 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
Keywords: CBSST; Schizoaffective Disorder; Psychotic Disorder; Cognitive Behavioral Therapy; Social Skills Training; Assertive Community Treatment
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Community Mental Health Services

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT + CBSST (Experimental): Implementing Cognitive Behavioral Social Skills Training in an Assertive Community Treatment model
  Interventions: Behavioral: Cognitive Behavioral Social Skills Training (CBSST)
- ACT only (Active Comparator): Assertive Community Treatment only
  Interventions: Other: Assertive Community Treatment (ACT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Social Skills Training (CBSST) — CBSST integrates CBT and SST techniques and neurocognitive compensatory aids. The treatment manual includes a patient workbook that describes the skills and includes homework assignment forms. Cognitive therapy is combined with role play practice of communication skills and problem-solving training. The ACT-adapted, team-delivered individual CBSST intervention will be delivered in 3 6-session modules (Cognitive Skills, Social Skills, and Problem Solving Skills) for a total of 18 weekly individual therapy sessions, but with participants completing the sequence of 3 modules twice, for a total of 36 sessions (9 months).
  Other Names: CBT; SST
  Arms: ACT + CBSST
Other: Assertive Community Treatment (ACT) — Assertive Community Treatment model is a evidence based practice model. ACT teams are multi-disciplinary and provide comprehensive services to individuals in their natural setting with small staff to recipient ratio. ACT teams use assertive engagement to proactively engage individuals in treatment providing services and support directly to individuals that are tailored to meet their specific goals and needs.
  Other Names: ACT
  Arms: ACT only

SUMMARY:
This project is an effectiveness trial comparing two psychosocial treatments for schizophrenia: Assertive Community Treatment (ACT) + Cognitive Behavioral Social Skills Training (CBSST) v. ACT, alone.

DETAILED DESCRIPTION:
Assertive community treatment (ACT) is one of the most well-validated treatment models for people with severe mental illness, and ACT is one of the few evidence-based practices that is widely implemented in community mental health programs; however, existing ACT approaches have little impact on functioning. The ACT model provides a unique opportunity for implementation of recovery-oriented EBPs throughout community mental health programs in the US. This project will examine the incremental effectiveness of implementing cognitive-behavioral strategies and social skills training in ACT relative to ACT, alone. The investigators will begin to examine a potential mechanism of change involving defeatist performance beliefs that can interfere with performance of community functioning behaviors, and will use qualitative methods to identify barriers and factors that contribute to successful implementation.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-diagnosis of schizophrenia or schizoaffective disorder at any stage of illness

Exclusion Criteria:

* Unstable assignment (at least 3 months) to an ACT team;
* Prior exposure to SST or CBT in the past 5 years
* Level of care required interferes with outpatient therapy (e.g., current hospitalization for psychiatric, substance use or physical illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2012-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Independent Living Skills Survey (ILSS) | Baseline, 18 mos.
  The ILSS is 70 item self-report measure in an interview format to assess everyday functioning. Each item is rated from 0 (No) to 1 (Yes). Scales are summed to yield a total score. Higher scores represent a higher level of functioning.

SECONDARY OUTCOMES:
Expanded Brief Psychiatric Rating Scale (BPRS) - Positive symptom factor structure | Baseline, 18 mos.
  The expanded BPRS is a 24-item scale that measures psychiatric symptom severity. Each item is rated from 1 (not reported) to 7 (very severe). Items are summed to yield a total factor score. Higher scores represent higher positive symptom severity.
Scale for Assessment of Negative Symptoms (SANS) | Baseline, 18 mos.
  The SANS is a 25 item semi-structured clinical interview designed to assess negative symptoms. The first 13 items measure diminished expression which consists of two domains: Affective flattening and Alogia. Each item is rated from 0 (Absent) to 5 (Severe). The total score is derived from the average of the Affective Flattening and Alogia global ratings (items #8 and #13)
Defeatist Performance Attitude Scale (DPAS) | Baseline, 18 mos.
  The DPAS is a 15-item self-report subscale of the commonly-used 40-item Dysfunctional Attitude Scale (DAS) used to measure generalized defeatist beliefs about one's ability to perform tasks and effectiveness of social behaviors. Each item is rated from 1 (agree completely) to 7 (disagree completely). Higher total scores (range = 15-105) indicate more severe defeatist performance attitudes.
Maryland Assessment of Social Competence (MASC) | Baseline, 18 mos.
  The MASC is a structured behavioral role play assessment that measures the ability to resolve interpersonal problems through conversation in three role play scenarios. Videotaped role plays are rated by blinded raters on three dimensions; verbal content, nonverbal communication behavior, and overall effectiveness, which will be the primary MASC variable. Each item is rated from 1 (very poor) to 5 (very good). A higher score for that dimension reflects higher ability and skills to solve problems in an interpersonal context.
Comprehensive Modules Test (CMT) | Baseline, 18 mos.
  The Comprehensive Module Test (CMT) is an assessment of CBSST skills acquisition. Scores are summed to yield a total CMT score range from 0-33. Higher total scores represent higher level of CBSST skills acquisition.
Cognitive Therapy Scale for Psychosis (CTS-Psy) | Baseline, 18 mos
  The Cognitive Therapy Scale for Psychosis (CTS-Psy) is 10 item scale for assessing the quality of cognitive behavior therapy. Items are scored on a scale from 0 to 6, where the total maximum achievable is 60. Higher scores indicate greater level of competency.
Dartmouth Assertive Community Treatment Scale (DACTS) | Baseline, 18 mos
  The DACTS is an assessment of assertive community treatment service fidelity. It consists of 28 items, each rated on a behaviorally-anchored scale from 1(not implemented) to 5 (fully implemented). The mean score for the total scale will be used as the measure of ACT team fidelity. A DACTS score of >4.0 is considered moderately high fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Granholm, PhD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wykes T, Steel C, Everitt B, Tarrier N. Cognitive behavior therapy for schizophrenia: effect sizes, clinical models, and methodological rigor. Schizophr Bull. 2008 May;34(3):523-37. doi: 10.1093/schbul/sbm114. Epub 2007 Oct 25. PMID 17962231
- [Background] Kurtz MM, Mueser KT. A meta-analysis of controlled research on social skills training for schizophrenia. J Consult Clin Psychol. 2008 Jun;76(3):491-504. doi: 10.1037/0022-006X.76.3.491. PMID 18540742
- [Background] Granholm E, McQuaid JR, McClure FS, Auslander LA, Perivoliotis D, Pedrelli P, Patterson T, Jeste DV. A randomized, controlled trial of cognitive behavioral social skills training for middle-aged and older outpatients with chronic schizophrenia. Am J Psychiatry. 2005 Mar;162(3):520-9. doi: 10.1176/appi.ajp.162.3.520. PMID 15741469
- [Background] Granholm E, McQuaid JR, McClure FS, Link PC, Perivoliotis D, Gottlieb JD, Patterson TL, Jeste DV. Randomized controlled trial of cognitive behavioral social skills training for older people with schizophrenia: 12-month follow-up. J Clin Psychiatry. 2007 May;68(5):730-7. doi: 10.4088/jcp.v68n0510. PMID 17503982
- [Background] Aarons GA, Wells RS, Zagursky K, Fettes DL, Palinkas LA. Implementing evidence-based practice in community mental health agencies: a multiple stakeholder analysis. Am J Public Health. 2009 Nov;99(11):2087-95. doi: 10.2105/AJPH.2009.161711. Epub 2009 Sep 17. PMID 19762654
- [Derived] Pillny M, Mueser KT, Holden J, Aarons GA, Sommerfeld D, Perivoliotis D, Granholm E. Enhancing Assertive Community Treatment With Cognitive Behavioral Social Skills Training for Schizophrenia: II. Ecological Momentary Assessment Outcomes in a Pragmatic Randomized-Controlled Trial. Schizophr Bull. 2025 Dec 14:sbaf103. doi: 10.1093/schbul/sbaf103. Online ahead of print. PMID 41391109
- [Derived] Granholm E, Mueser KT, Holden JL, Worley M, Sommerfeld D, Perivoliotis D, Ehret B, Pillny M, Aarons GA. Enhancing Assertive Community Treatment with Cognitive Behavioral Social Skills Training for Schizophrenia: I. Primary Outcomes in a Pragmatic Randomized-Controlled Trial. Schizophr Bull. 2025 Dec 14:sbaf084. doi: 10.1093/schbul/sbaf084. Online ahead of print. PMID 41391103
- [Derived] Sommerfeld DH, Aarons GA, Naqvi JB, Holden J, Perivoliotis D, Mueser KT, Granholm E. Stakeholder Perspectives on Implementing Cognitive Behavioral Social Skills Training on Assertive Community Treatment Teams. Adm Policy Ment Health. 2019 Mar;46(2):188-199. doi: 10.1007/s10488-018-0904-8. PMID 30406858
- [Derived] Granholm E, Holden JL, Sommerfeld D, Rufener C, Perivoliotis D, Mueser K, Aarons GA. Enhancing assertive community treatment with cognitive behavioral social skills training for schizophrenia: study protocol for a randomized controlled trial. Trials. 2015 Sep 30;16:438. doi: 10.1186/s13063-015-0967-8. PMID 26424639